CLINICAL TRIAL: NCT03175770
Title: Feasibility of Radiofrequency Resection in Oropharyngeal Tumor Surgery
Status: Completed | Type: Observational
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Other Study IDs: 381/14
Record Dates: First submitted 2017-03-16; First posted 2017-06-05 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Radiofrequency Resection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with benign or malign tumor in the oropharynx: Patient of 18 years and older with benign or malign tumor in the oropharynx. The resection is done transorally by radiofrequency
  Interventions: Procedure: transoral radiofrequency Resection in Oropharyngeal Tumor Surgery

INTERVENTIONS:
Procedure: transoral radiofrequency Resection in Oropharyngeal Tumor Surgery — Patient of 18 years and older with benign or malign tumor in the oropharynx. The resection is done transorally by radiofrequency

SUMMARY:
In the last years radiofrequency resection has become a frequent method in surgical subspecialties. Although many departments are using this method for the resection of Tumor in the oropharynx, there is no study so far which describes feasibility and safety.

Goal of this study is to show feasibility and safety of Radiofrequency Resection in Oropharyngeal Tumor Surgery.

DETAILED DESCRIPTION:
In the last years radiofrequency resection has become a frequent method in surgical subspecialties. Although many departments are using this method for the resection of Tumor in the oropharynx, there is no study so far which describes feasibility and safety.

Goal of this study is to show feasibility and safety of Radiofrequency Resection in Oropharyngeal Tumor Surgery.

ELIGIBILITY:
Inclusion Criteria:

- 18 years and older benign or malign tumor of the oropharynx tumor must be resectable transorally

Exclusion Criteria:

* Prior radiotherapy or chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 18 years or older, benign or malign tumor of the oropharynx. the resection must be done transorally
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-15 (Actual)

PRIMARY OUTCOMES:
total blood loss, | intraoperative
  assessing the blood loss by measuring blood in the suction
tissuesticking | intraoperative
  tissuesticking by physician global assessment scale from 1 - 6
coagulation | intraoperative
  coagulation by physician global assessment scale from 1 - 6,
Duration of Operation | intraoperative
  measuring Duration of Operation in minutes

SECONDARY OUTCOMES:
Zone of coagulation | within one month after the operation
  Zone of coagulation to assess the tissue damage by radiofrequency by a scale 1 - 6,
postoperative parameters | within one month after the operations
  woundhealing by Parameters normal, delayed, infection;
postoperative pain | within one month after the operations
  postoperative pain by visual analog scale from 0 -10,
accuracy of section | within one month after the operations
  accuracy of section assessed by a scale from 1 - 6
status of resection | within one month after the operations
  assessment of status of resection by assessing the margins of resection for Tumor scale from 1 - 6,
postoperative dysfunctions by descriptive name of scale | within one month after the operations
  postoperative dysfunctions by descriptive scale from 1 -10

CONTACTS AND LOCATIONS:
Overall Officials: Clemens Heiser, MD, Principal Investigator — department for ENT, Klinikum Rechts der Isar der Technischen Universität München, Ismaninger Straße 22, 81675 München, Germany
Locations (1):
- Department of Ear Nose Throat, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researchers